CLINICAL TRIAL: NCT03442075
Title: Prospective, Controlled, Randomized Clinical Trial to Evaluate the Effectiveness of Four Analgesic Methods During Trans Rectal Prostate Biopsy.
Brief Title: Pain Comparison Whit Visual Analog Scale (EVA) Between Four Analgesic Methods During Trans Rectal Prostatic Biopsy
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, EDGAR BELTRAN-SUAREZ, Dr Edgar Beltran-Suarez, Instituto Mexicano del Seguro Social
Other Study IDs: R-2017-3501-61
Record Dates: First submitted 2018-02-10; First posted 2018-02-22 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Cancer of Prostate
Keywords: Cancer of Prostate; Analgesic method
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Group 1 an analgesic suppository was applied
- Group 2: Group 2 was administered analgesic orally
- Group 3: Group 3 was given trans rectal gel
- Group 4: Group was performed peri prostatic infiltration.
- Group 5: Group was performed by placebo oral

SUMMARY:
Define the best analgesic method between peri prostatic blockage, analgesic suppository, oral analgesic and topic anesthetic gel, during trans rectal prostate biopsy

DETAILED DESCRIPTION:
Comparison between four analgesic methods during trans rectal prostatic biopsy.

OBJECTIVE: To define the best analgesic method between the peri-prostatic block, the analgesic suppository, the oral analgesic, the final anesthetic gel, during the trans rectal prostate biopsy determined at the end of the procedure with a visual analogue scale for pain (VAS pain) in a Interview 15 to 30 minutes at the end of the procedure.

METHODS: experimental, retrospective, longitudinal, comparative, during May to July 2017, 350 trans rectal prostate biopsies were performed, all cases were randomly assigned to one of the four study groups. The data analysis will be performed by calculating measures of central tendency and dispersion for quantitative variables and ANOVA test, for qualitative variables Chi square to determine statistical differences between the three moments of pain in the parameters of introduction of the ultrasound transducer, sampling of Prostate of the minimum 12 biopsies and discomfort in general of the procedure

ELIGIBILITY:
Inclusion Criteria:

* Male patients older than 18 years with indication for trans rectal prostate biopsy

Exclusion Criteria:

* Bad intestinal preparation.
* Painful anorectal pathologies.
* Clotting disorders without previous assessment by hematology.
* Acute prostatitis

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The patients from the consultation were taken from the first time they were derived from the peripheral clinics or from the ones derived from our same medicine, with suspicion of prostate cancer and that the criteria for carrying out the trans rectal prostate biopsy were met.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Ultrasound Transducer | Interview 15 to 30 minutes at the end of the procedure
  Evaluation of the discomfort or pain in the introduction of the trans rectal ultrasound transducer determined at the end of the procedure with Visual Analog Scale for Pain, which is a psychometric measuring instrument designed to assess the pain intensity experienced by each patient individually. Was employ for first time in 1921 and referred as a "graphical rating method", which has the characteristic of being able to achieve a rapid classification (statistically measurable and reproducible) of the severity of pain experience.
  The analogous visual scale used for this study measures from 0-10 the intensity of the pain with a series of "faces" that show the intensity in the pain experimentation with categories like "No pain" approximately 0-1, mild, annoying in number 2, nagging in number 4, distressing in number 6, intense in number 8 and worst possible in number 10.

SECONDARY OUTCOMES:
Biopsy | Interview 15 to 30 minutes at the end of the procedure
  Evaluation of the discomfort or pain at the moment of the biopsy, that is, when the needle is inserted to take the samples in a 12-cylinder minimum or as needed, determined at the end of the procedure with Visual Analog Scale for Pain, The analogous visual scale used for this study measures from 0 to 10 the intensity of pain with a series of "faces" that show the intensity in the pain experimentation with categories such as "No pain" approximately 0-1, mild, annoying in number 2, annoying in number 4, distressing in number 6, intense in number 8 and worse in number 10.
  The analogous visual scale used for this study measures from 0-10 the intensity of the pain with a series of "faces" that show the intensity in the pain experimentation with categories like "No pain" approximately 0-1, mild, annoying in number 2, nagging in number 4, distressing in number 6, intense in number 8 and worst possible in number 10.

OTHER OUTCOMES:
General procedure | Interview 15 to 30 minutes at the end of the procedure
  Evaluation of the discomfort or pain at the moment of the biopsy, that is, when the needle is inserted to take the samples in a 12-cylinder minimum or as needed, determined at the end of the procedure with Visual Analog Scale for Pain. The analogous visual scale used for this study measures from 0 to 10 the intensity of pain with a series of "faces" that show the intensity in the pain experimentation with categories such as "No pain" approximately 0-1, mild, annoying in number 2, annoying in number 4, distressing in number 6, intense in number 8 and worse in number 10.

CONTACTS AND LOCATIONS:
Overall Officials: EDGAR BELTRAN-SUAREZ, MD, Principal Investigator — HOSPITAL OF SPECIALTIES OF THE NATIONAL MEDICAL
Locations (1):
- Edgar Beltran-Suarez, Mexico City, Aztcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Attard G, Parker C, Eeles RA, Schroder F, Tomlins SA, Tannock I, Drake CG, de Bono JS. Prostate cancer. Lancet. 2016 Jan 2;387(10013):70-82. doi: 10.1016/S0140-6736(14)61947-4. Epub 2015 Jun 11. PMID 26074382
- [Background] Lowrance WT, Roth BJ, Kirkby E, Murad MH, Cookson MS. Castration-Resistant Prostate Cancer: AUA Guideline Amendment 2015. J Urol. 2016 May;195(5):1444-1452. doi: 10.1016/j.juro.2015.10.086. Epub 2015 Oct 20. PMID 26498056
- [Background] Loeb S, Vellekoop A, Ahmed HU, Catto J, Emberton M, Nam R, Rosario DJ, Scattoni V, Lotan Y. Systematic review of complications of prostate biopsy. Eur Urol. 2013 Dec;64(6):876-92. doi: 10.1016/j.eururo.2013.05.049. Epub 2013 Jun 4. PMID 23787356
- [Background] Mottet N, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Schmid HP, van der Kwast T, Wiegel T, Zattoni F, Heidenreich A. [EAU guidelines on prostate cancer. Part II: treatment of advanced, relapsing, and castration-resistant prostate cancer]. Actas Urol Esp. 2011 Nov-Dec;35(10):565-79. doi: 10.1016/j.acuro.2011.03.011. Epub 2011 Jul 14. Spanish. PMID 21757258
- [Background] Herranz Amo F, Diez Cordero JM, Cabello Benavente R. [Evolution of the transrectal ultrasound guided prostatic biopsy technique]. Arch Esp Urol. 2006 May;59(4):385-96. Spanish. PMID 16800136
- [Background] Sahin A, Ceylan C, Gazel E, Odabas O. Three different anesthesia techniques for a comfortable prostate biopsy. Urol Ann. 2015 Jul-Sep;7(3):339-44. doi: 10.4103/0974-7796.152014. PMID 26229322
- See also: National Cancer Institute. A Snapshot of Prostate Cancer: Incidence and Mortality — http://www.cancer.gov/research/progress/snapshots/prostate
- See also: WHO | GLOBOCAN 2012 Estimated Cancer Incidence, Mortality and Prevalence Worlwide in 2012 [Internet]. 2015 [cited 2016 Mar 21]. p. 3. Available from: — http://globocan.iarc.fr/Pages/fact_sheets_population.aspx